CLINICAL TRIAL: NCT06901843
Title: Comparative Effects of Closed Kinetic Chain Exercises and Mobilization Exercises in Elderly Females With Neck of Femur Fracture
Brief Title: Comparative Effects of Closed Kinetic Chain Exercises and Mobilization Exercises in Elderly Females With NFF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/778
Record Dates: First submitted 2025-03-23; First posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Neck of Femur Fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobilizations Exercises (Experimental)
  Interventions: Combination Product: Mobilizations Exercises
- Closed Kinetic Chain Exercises (Active Comparator)
  Interventions: Combination Product: Closed Kinetic Chain Exercises

INTERVENTIONS:
Combination Product: Mobilizations Exercises — Group A was treated with mobilizations exercises for 40 minutes for 3 sessions per week for 6 weeks. Patients received hip mobilizations. Therapist perform anterior posterior glide, caudal glide, posterior anterior glide with abduction, flexion and lateral rotation in 3 sets with 10 repetitions .Mobilization grades were performed according to patients tolerance level with duration 30-second rest .Hip strengthening exercises were performed 3 sets with 10 repetition with hip abduction in side lying, hip extension in prone position, sideway walk, hip abduction in a stand up position.
  Arms: Mobilizations Exercises
Combination Product: Closed Kinetic Chain Exercises — Group B was treated with Closed Kinetic Chain Exercises for 40 minutes for 3 sessions per week for 6 weeks. Closed kinetic chain exercises were performed with 5 minute break between each exercise. Leg press in horizontal position ,Stationary bicycling and Stairmaster climbing.
  Arms: Closed Kinetic Chain Exercises

SUMMARY:
This study investigates the additional benefits of Mobilization Exercises and Closed Kinetic Chain Exercises (CKCE) in elderly individuals with post-operative neck of femur fracture. The researcher employs a randomized controlled trial which will involve 49 participants aged above 65 years with post-operative neck of femur fracture.

DETAILED DESCRIPTION:
Participants are divided into two groups:

one receiving Mobilization Exercises, and the other receiving Closed Kinetic Chain Exercises. Outcomes are assessed over a 6 week period, focusing on pain intensity, Range of motion, risk of fall by goniometer, visual analogue scale (VAS) and dynamic gait index (DGI) scores. Data will be analyzed using SPSS-23. The study will conclude whether CKCE or Mobilization exercises offer a significant benefit in pain reduction, prevent risk of falls and range of motion.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by Orthopedic Surgeon with neck of femur fracture by x ray findings
* Patients undergone surgical treatment for neck of femur fracture within one year.
* Patients administer in groups after 12 weeks of post-operative period
* X-ray reexamination with no fracture or dislocation before treatment
* Ability to walk normally or with crutches
* Patients walk without any assistance before injury
* Un-displaced neck of femur fracture according to Garden Classification
* Operated on using internal fixation
* Only females were included
* Aged 65 years or older

Exclusion Criteria:

* Bilateral hip fracture
* Bedridden patient before fracture
* Patient who have undergone any previous surgery of lower limb
* Neurological Condition

Min Age: 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-03-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | 12 Months
  The 10-point numeric scale ranges from '0' representing "no pain" to '10' representing "pain as bad as you can imagine" or "worst pain imaginable". The VAS is a valid and reliable scale to measure pain intensity. VAS demonstrates strong correlation validity with other established pain measurement scales, making it a reliable tool for clinical assessments. Validity is 0.88 % and Reliability is 0.90%.
Dynamic Gait Index (DGI) | 12 months
  The questionnaire has been designed to evaluate risk of fall and balance during dynamic tasks. DGI includes 8 items, score between 0-3 scales. Score of 0 indicates severe impairment and score of 3 indicates normal function. Total score is between 0-24. Validity is 0.88% and Reliability is 0.97%. Interpretation 0-11: Severe impairment 12-19: Moderate impairment 20-24: Mild impairment
GONIOMETER | 12 months
  Goniometer is used to measure the joint angle in degrees, ROM and flexibility. The goniometer measures ranges and degrees of joints. The range of goniometer is typically 0-180 degrees or o-360 degrees. The intervals on scale can vary from 0-10 degrees. Hip Joint Ranges of Motion
  1. Flexion: 120-130 degrees
  2. Extension: 10-20 degrees
  3. Abduction: 40-50 degrees
  4. Adduction: 20-30 degrees
  5. Internal Rotation: 30-40 degrees
  6. External Rotation: 40-50 degrees

CONTACTS AND LOCATIONS:
Locations (1):
- Bajwa hospital J7JP+4WH, GT Rd, Shahdara Town, Shahdara, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No